CLINICAL TRIAL: NCT02791711
Title: Using Nasal Broadband Glasses HFNC (High Flow Nasal Cannula) in the Initial Management of Severe Bronchiolitis in Infants Admitted in ICU: Bicentric Observational Study on the 2013-2014 Epidemic
Brief Title: Using Nasal Broadband Glasses in the Initial Management of Severe Bronchiolitis in Infants Admitted in ICU
Acronym: HFNC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 14-HPNCL-09
Record Dates: First submitted 2016-06-01; First posted 2016-06-07 (Estimated); Last update posted 2019-08-01 (Actual); Status verified 2016-06

CONDITIONS: Bronchiolitis
Keywords: Bronchiolitis; Continuous Positive Airway Pressure; HFNC
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- High Flow Nasal Cannula (Other): Use of High Flow Nasal Cannula
  Interventions: Other: High Flow Nasal Cannula

INTERVENTIONS:
Other: High Flow Nasal Cannula — Evaluation of the use of High Flow Nasal Cannula by biological markers, questionary of quality of use of HFNC by the physician, questionary of evaluation of adverse events with HFNC

SUMMARY:
The aim of this study is to evaluate the use of nasal broadband glasses HFNC (High Flow Nasal Cannula) in the initial management of severe bronchiolitis in infants admitted in ICU.

Nasal HFNC can deliver warmed humidified gas through a nasal interface, greatly improving the safety and efficacy of administering O2. This device generates a continuous positive pressure in the airways, to reduce the work of breathing. The sealing absence of the HFNC at the nasal interface improves patient comfort and avoiding nasal trauma.

DETAILED DESCRIPTION:
Bronchiolitis in infants is a common and potentially serious disease. It corresponds to an acute pulmonary disease and dyspnea usually viral (70 to 80% of Respiratory syncytial virus (RSV) in infants less than 1 year). It particularly affects infants under 2 years.

The 2001 consensus conference and bronchiolitis 2006 on the management clarified the criteria for hospitalization and simplified therapeutic attitudes. These conferences have highlighted the importance of humidification, the nasopharyngeal desobstruction for less severe forms of oxygen therapy and for others. Recent literature has also shown that the use of noninvasive ventilation type Continuous Positive Airway Pressure (CPAP) nasal or broadband nasal glasses (HFNC: High Flow Nasal canula) in severe forms possible to reduce the work of breathing of children with severe bronchiolitis and their use in studies "before / after" was accompanied by a significant decrease in the use of invasive ventilation.

The HFNC and nasal CPAP can deliver warmed humidified gas through a nasal interface, greatly improving the safety and efficacy of administering O2. These devices generate a continuous positive pressure in the airways, for decreasing the work of breathing. The sealing absence of the HFNC at the nasal interface improves patient comfort and avoiding nasal trauma, sometimes encountered with nasal CPAP interfaces.

The HFNC is a simple, effective and safe, commonly used in severe bronchiolitis admitted in ICU (Intensive Care Unit). However instead of this technique is not yet well defined.

The investigators assume that the use of HFNC in severe bronchiolitis in first line allows sufficient respiratory improvement to avoid recourse to other technical assistance ventilatory more binding.

ELIGIBILITY:
Inclusion Criteria:

* In which the diagnosis of bronchiolitis is strongly suspected (1st or nth episode). Acute bronchiolitis is defined by the presence of respiratory distress (wheezing, crackles auscultatory, wrestling signs) or apnea can not be explained by another existing pathology in children with a clinical history of upper respiratory infection.
* Satisfactory at least 1 of the following severity criteria:

EN> 50 quiet,

* Trouble consciousness / hypotonia,
* Significant Apnea (with desaturation and / or bradycardia)
* Hypercapnic acidosis (pH <7.3 and carbon dioxide partial pressure (PCO2)> 55mmHg)
* Oxygen saturation (SpO2) <92% on room air
* Including the holders of parental authority / legal representative are informed of the study and expressed no opposition to the participation of their child.
* Affiliated with a social security scheme by one of the holders of parental authority / legal guardian

Exclusion Criteria:

* Children with neuromuscular disease known heart or lung (even without decompensation) at the time of admission.
* Any vital distress, including respiratory or neurological justifying intubation or other emergency resuscitation gesture.
* Opposition to a parent / guardian to the participation of their children in the study.
* Desire to study withdrawal expressed by one of the holders of parental authority / legal guardian
* Voluntary or involuntary break current care protocol or research by the healthcare team.

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2013-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Rate of early success for the number of bronchiolitis who once admitted in the ICU and placed HFNC will not need another support ventilation mode after one hour of treatment (H1) | after one hour of treatment
  the number of children who once set HFNC at baseline Hour 0 will not need another breathing assistance technique After 1 hour H1 of treatment

SECONDARY OUTCOMES:
Overall success rate | Comparison between baseline Hour 0 and after 1 hour of treatment
  Number of children who will not need another technique while respiratory assistance throughout the ICU stay
Demographic predictive factors of failure of HFNC | At baseline hour 0
  Correlation of demographic data Hour 0 to failure of HFNC
Clinical predictive factors of failure of HFNC | At baseline hour 0
  Correlation of clinical data Hour 0 to failure of HFNC
The child's comfort HFNC | comparison to Hour 0, Hour 1, Hour 12
  Neonatal pain and discomfort scale " Échelle Douleur Inconfort Nouveau-Né" (EDIN)) Scores comparison to Hour 0, Hour 1, Hour 12
  This scale evaluates the prolonged pain and discomfort of the child, an hetero assesor measures by 5 items about face, body, sleep, comfort and relationship. Each item scores from 0 to 5. 0 means no pain or discomfort symptoms and 5 means the maximum symptoms.
  Global score will be from 0 to 15.
Incidence of adverse events in HFNC | From baseline hour 0 to the end of hospitalization
  Frequency and types of adverse events throughout the ICU hospitalization period
Effectiveness of HFNC after 1 hour of application | Comparison between baseline Hour 0 and after 1 hour of treatment
  comparaison of clinical data between baseline and 1 Hour of HFNC application.

CONTACTS AND LOCATIONS:
Overall Officials: Mickael AFANETTI, MD, Principal Investigator — Fondation LENVAL - Hôpitaux Pédiatriques de Nice CHU-LENVAL
Locations (2):
- France (2):
  - Hôpital Arnaud de Villeneuve - CHU de Montpellier, Montpellier
  - Fondation LENVAL - Hôpitaux Pédiatriques de Nice CHU-LENVAL, Nice

IPD SHARING:
Plan to Share IPD: No